CLINICAL TRIAL: NCT02942173
Title: A Phase II Prospective Randomized Trial of Donor T-memory Cells (CD45RA Depleted) Infusion for Prevention of Infections After Allogeneic TcRαβ/CD19-depleted Hematopoietic Stem Cell Transplantation
Brief Title: CD45RA Depleted T-cell Infusion for Prevention of Infections After TCRab/CD19-depleted Allo-HSCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CD45RAndom_2016_1
Record Dates: First submitted 2016-10-11; First posted 2016-10-21 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; GvHD; Opportunistic Infections; Graft-versus-Host Disease
Keywords: CD45RA-depletion; TCR-alpha/beta depletion; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Opportunistic Infections; Graft vs Host Disease

ARMS (2):
- CD45RA- (No Intervention)
- CD45RA+ (Experimental)
  Interventions: Biological: CD45RA-depleted peripheral blood mononuclear cells

INTERVENTIONS:
Biological: CD45RA-depleted peripheral blood mononuclear cells — Infusion of escalating doses of CD45RA-depleted donor-derived allogeneic peripheral blood mononuclear cells
  Arms: CD45RA+

SUMMARY:
The purpose of this prospective randomized study is to determine whether infusions of T-memory cells prevent infections in children with leukemia after allogeneic alpha, beta T-cell receptor (TcRab)/CD19-depleted hematopoietic stem cell transplantation (HSCT).

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) remains the most important direct complication of hematopoietic stem cell transplantation. Methods used to prevent GVHD include diverse pharmacologic interventions and ex vivo methods of T-cell depletion, the latter being the most effective ones. Historically depletion of T-cells from the graft is associated with increased rate of graft failure, relapse of malignant disease and prolonged immune deficiency. Selective depletion of TCR-alpha/beta T-lymphocytes is a new method of hematopoietic stem cell graft manipulation, which is thought to conserve important cell populations, e.g. NK cells and gamma/delta T cells within the graft. Preliminary results suggest that TCR alpha/beta depletion ensures high engraftment rate, low early mortality and good control of GVHD. The problem of delayed immune reconstitution and life-threatening viral infections remains incompletely resolved.

Depletion of naive (CD45RA-positive) T-cells was developed as a new method of graft manipulation to prevent GVHD. Research data indicate that alloreactivity is associated mainly with naive T-cell fraction. In vitro depletion of CD45RA lowers significantly the alloreactive response while retaining reactivity to pathogens.

In previous pilot protocol the investigators confirmed that infusion after TCR-alpha/beta depleted transplantation of low doses of CD45RA-depleted mononuclear cells are safe and potentially protective against viral infections. The biologic readout for the protocol was a quantitative assessment of T-cell reactivity to common pathogens after infusion and owing to the trial results expansion of CMV-specific CD8 T-cells was discovered in most of the patients.

In current randomized protocol the investigators are posing a question if donor lymphocytes infusion (DLI) of low doses of CD45RA-depleted mononuclear cells are effective in viral prophylaxis after TCR-alpha/beta depleted transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered candidates for allogeneic hematopoietic stem cell transplantation and have one of the following diagnoses:

  * Acute lymphocytic leukemia (ALL)
  * Acute myeloid leukemia
  * Acute biphenotypic leukemia
  * Acute bilinear leukemia
  * Lymphoma
  * Myelodysplastic syndrome
  * Chronic myeloid leukemia
* Transplant processing: TCR ab/CD19-depletion
* Donors:

  * HLA-match unrelated volunteers
  * Partly and haploidentical relative

Exclusion Criteria:

* ALL patients not in remission
* Patients with uncontrolled infections
* Clearance of creatinine < 70 ml/min
* Cardiac ejection fraction < 40%
* Patients who can perform pulmonary function tests will be excluded if they have a diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) of < 50% predicted; patients who are unable to perform pulmonary function tests will be excluded if the oxygen (O2) saturation is < 92% on room air
* Patients who have liver function test (LFTs) (including total bilirubin, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) >= twice the upper limit of normal
* Mental disease of both patient, patient's tutor (if patient is under age 18) and donor, that hinder understanding of main point of the study and keeping treatment plan, hygiene and sanitation

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of the probability of CMV-reactivation after HSCT | 120 days after HSCT
cumulative incidence of acute GVHD grade II-IV. | 150 days after HSCT

SECONDARY OUTCOMES:
cumulative incidence of of CMV-disease at 100,180 and 365 days after HSCT | 100, 180 and 365 days after HSCT
overall survival at 365 days after HSCT | 365 days after HSCT
Event-free survival at 365 days after HSCT | 365 days after HSCT
cumulative incidence of relapse at 6 months and 365 days after HSCT | 6 months and 365 days
cumulative incidence of transplant-related mortality at 6 months after HSCT | 6 months
cumulative incidence of chronic GvHD | 1 year after HSCT
cumulative incidence of neutrophil and platelets engraftment at 14 and 30 days after HSCT | 14 and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maschan, PhD, Study Director — Fedaral Research Center for pediatric hematology, oncology and immunology; Larisa Shelikhova, PhD, Study Chair — Fedaral Research Center for pediatric hematology, oncology and immunology
Locations (1):
- Federal Research Center for pediatric hematology, oncology and immunology, Moscow, Russia